CLINICAL TRIAL: NCT04298684
Title: Efficacy of Metformin Versus Sitagliptin on Benign Thyroid Nodules Size in Type 2 Diabetes: a 2-years Prospective Multicentric Study
Brief Title: Efficacy of Metformin Versus Sitagliptin on Benign Thyroid Nodules in Type 2 Diabetes
Acronym: METNODTHYR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PAP_RI1_2019/1; 2019-000676-42 (EudraCT Number)
Record Dates: First submitted 2020-02-05; First posted 2020-03-06 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 2; Thyroid Nodule (Benign)
Keywords: type 2 diabetes mellitus; thyroid nodule; metformin; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Thyroid Nodule; Insulin Resistance | interventions — Metformin; Sitagliptin Phosphate

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective open-label study evaluating the efficacy of metformin compared to sitagliptin on benign TN growth in subjects with T2DM. After written approval, subjects with T2DM who meet the eligibility criteria will have a thyroid ultrasound. Subjects with TN of at least 2 cm and 2 benign cytology results after fine-needle aspiration, will be included after a run-in period of 1 month with a daily basal insulin therapy in order to reduce glucotoxicity. If the Hb1Ac levels remain above 8%, the subjects will not be included. After inclusion, a central randomization will allow subjects to benefit from either metformin (group 1) or sitagliptin (group 2). In both cases, the standard nutritional care and physical activity recommendations (150 minutes of physical activity per week) will be recalled. If HbA1c levels > 8% during the follow-up, treatment by gliclazide will be introduce (LP30mg). A follow-up schedule will be given to the included patient for future visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): In arm 1, the subjects will receive metformin at the initial dose of 500mg x 2 / day, which will be increased weekly to 500mgx3 / day and then 1gx2 / day in order to obtain the minimum effective dose on glycemic control.
  Interventions: Drug: METFORMIN
- Sitagliptin (Placebo Comparator): In arm 2, sitagliptin will be prescribed at 100mg / day. A classic follow-up will be done every 3 months.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: METFORMIN — After inclusion, a central randomization will allow subjects to benefit from either metformin (group 1) or sitagliptin (group 2). A follow-up schedule will be given to the included patient for future visits. thyroid ultrasonography to analyze the TN evolution in the 2 groups.
  In arm 1, the subjects will receive metformin at the initial dose of 500mg x 2 / day, which will be increased weekly to 500mgx3 / day and then 1gx2 / day in order to obtain the minimum effective dose on glycemic control. In case of intolerance, the tolerated and effective dose will be taken back provided an effective glycemic control.
  A classic follow-up will be done every 3 months. Thyroid US and measure of HOMA-IR index will be done every 6 months for 2 years. If the goal of HbA1c will not achieved, a treatment with glicazide will be introduced.
  Arms: Metformin
Drug: Sitagliptin — After inclusion, a central randomization will allow subjects to benefit from either metformin (group 1) or sitagliptin (group 2). A follow-up schedule will be given to the included patient for future visits. thyroid ultrasonography to analyze the TN evolution in the 2 groups.
  In arm 2, sitagliptin will be prescribed at 100mg / day. A classic follow-up will be done every 3 months. Thyroid US and measure of HOMA-IR index will be done every 6 months for 2 years. If the goal of HbA1c will not achieved, a treatment with glicazide will be introduced.
  Arms: Sitagliptin

SUMMARY:
A 2-years prospective, randomized and multicentric study will be performed to assess the efficacy of metformin compared to sitagliptin on benign thyroid nodules size ≥ 2 cm, in newly diagnosed patients with type 2 diabetes.

DETAILED DESCRIPTION:
Previous studies reported that prevalence of thyroid nodules (TN) is increased in patients with insulin resistance (IR) and type 2 diabetes mellitus (T2DM). However, there are no guidelines for the management of TN in this target population. In 2013, the French National Health Insurance reported that thyroid surgery procedures for benign nodules have increased unjustifiably. The impact of such surgery on the patients could be serious, with psychological repercussions and risks of surgical complications and the need of a substitutive lifetime hormonal treatment. The investigators hypothesize that metformin may reduce the need of TN surgery by decreasing benign TN size through a reduction of IR profile. A 2-years multicentric prospective study will be conducted to compare efficacy of metformin versus sitagliptin on benign thyroid nodules size in patients with initial benign thyroid nodules ≥ 2 cm. The percentage of thyroid surgery avoided, IR profile measured by Homeostasis Model Assessment of Insulin Resistance-Index (HOMA-IR-index) and adipokines concentrations will be also collected at inclusion ad at 2 years. The Primary outcome will be the percentage of patients in each group who had at least a 20% decrease in one or more nodules of more than 2 cm at 2 years. Several secondary outcomes will be registered: percentage of thyroid surgery observed in each group at 2 years, number of new TN (≥ 10mm) after 2 years of follow-up , percentage of metabolic syndrome before and after treatment, proportion of subjects with improvement of the HOMA-IR index and adipokine concentrations, plasmatic thyroid-stimulating hormone (TSH), T4 and T3 levels evolution, percentage of insulin like growth factor-1 (IGF-1) and adiponectin receptor expression in thyroid tissues after TN surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM aged 18 to 65 years;
* Uncomplicated T2DM, evolving for less than 3 years;
* Patients with HbA1c levels between 7 and 8% (after the run-in period)
* Patients with at least one TN ≥ 2 cm non-cystic, whose benignity will be confirmed by a fine-needle aspiration cytology performed twice regardless of ultrasound TIRADS score;
* Naive subjects of any treatment: never received an anti-diabetic treatment OR received an anti-diabetic treatment of less than 30 days since diagnosis OR did not receive an anti-diabetic treatment during the 30 days before screening;
* Patients with a creatinine clearance > 60 ml/min;
* Informed and written consent signed by the patient and the investigator;
* Affiliation to the national social health system or equivalent.

Exclusion Criteria:

* Subjects without adequate or impaired decisional abilities for consent to research and placed under guardianship, trusteeship or safeguard of justice
* Pregnant or breastfeeding woman
* Woman of childbearing potential without effective contraception (estroprogestative, presentative, intrauterine device)
* Suspect thyroid nodules in ultrasound (TIRADS 4 to 5) with confirmation after a fine-needle aspiration cytology;
* Thyroid function abnormalities or a history of thyroid disease;
* Thyroid nodules whose size or symptoms (compressive signs) require surgery
* Ioduria <100ug /L
* Thyroid autoimmunity: positive anti-peroxidase, thyroglobulin or anti-TSH receptors antibodies
* Levothyroxine treatment
* History of cervical radiotherapy or thyroid surgery
* Type 1 diabetes
* Insulin deficiency
* History of hypersensitivity to one of the active substances
* History of pancreatitis
* Obesity linked to endocrine disease
* Presence of severe complications of T2DM (ischemic heart disease, heart failure with reduced left ventricular ejection fraction, severe lower extremity arteritis, gangrene, retinopathy, end-stage renal failure, cerebrovascular accident)
* HbA1c levels > 8% after the run-in period
* Liver diseases (liver failure, cirrhosis, viral hepatitis B or C)
* Acute alcoholic intoxication, chronic alcoholism
* Psychiatric diseases (depression, schizophrenia)
* Neurological diseases (epilepsy, demyelinating diseases, etc.)
* Treatment influencing the morphology or thyroid function: corticosteroids, lithium, iodized products etc. ...
* Acute conditions that may impair renal function such as: dehydration, severe infection, shock
* Respiratory failure
* Metabolic acidosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in each group who had at least a 20% decrease in one or more nodules of more than 2 cm at 2 years. | 24 months
  Size : The reduction of TN will be evaluated by thyroid ultrasonography. The operator will be the same throughout the follow-up and in each center, with an evaluation every 6 months. A measurement and precise analysis of the TN will be performed. If a TIRADS 4 or 5 classification is described , a new fine-needle aspiration cytology will be performed. A final thyroid ultrasonography evaluation will be performed at 2 years in order to allow the comparison of TN sizes from the pre-inclusion period to the final period.

SECONDARY OUTCOMES:
Percentage of thyroid surgery observed in each group at 2 years. | 24 months after treatment initiation
  Record the number of thyroid surgeries performed after inclusion for 2 years
Number of new TN (≥ 10mm) after 2 years of follow-up | Baseline and 24 months after treatment initiation
  Detection of new TN (≥ 10mm) by thyroid ultrasonography. The operator will be the same throughout the follow-up and in each center
Change between percentage of metabolic syndrome before and after treatment according to the NCEP ATP III definition | Baseline, every 6 months after treatment initiation until 24 months
  Central or abdominal obesity (measured by waist circumference):
  * Men - greater than 40 inches (102 cm)
  * Women - greater than 35 inches (88cm) Triglycerides plasmatic levels greater than or equal to 150 mg/dL (1.7 mmol/L)
  HDL cholesterol :
  * Men - Less than 40 mg/dL (1.03 mmol/L)
  * Women - Less than 50 mg/dL (1.29 mmol/L) Blood pressure greater than or equal to 130/85 mm Hg Fasting glucose greater than or equal to 110 mg/dL (6.1 mmol/L)
Proportion of subjects with improvement of the HOMA-IR index | Baseline, every 6 months after treatment initiation until 24 months
  The HOMA index will be measured after calculation the ratio between the [fasting plasma insulin (Mu / L) X Fasting plasma glucose (mmol / l)] / 22.5
Proportion of subjects with improvement of adipokine concentrations | Baseline and 24 months after treatment initiation
  Among the adipokines, we will measure the plasmatic Leptin, Adiponectin and Vifastin levels
Plasmatic thyroid hormon levels | Baseline, every 6 months after treatment initiation until 24 months
  these dosages will allow us to evaluate the changes in the functioning of the nodular thyroid gland during follow-up under either treatment
Percentage of IGF-1 receptor expression in thyroid tissues after TN surgery | through study completion, an average of 1 year
  The analysis of the tissue expression of IGF1 receptors will be performed on thyroid samples after surgery if performed. One sample will be frozen and another will be included in paraffin for further analysis. IGF1 receptors are involved in the insulin and glucose metabolism signaling pathways. Analysis of their expression could help us to understand the possible links between insulin resistance and thyroid nodule.
Percentage of adiponectin receptor expression in thyroid tissues after TN surgery | through study completion, an average of 1 year
  The analysis of the tissue expression of adiponectin receptor will be performed on thyroid samples after surgery if performed. One sample will be frozen and another will be included in paraffin for further analysis. Adiponectin receptor are involved in the insulin and glucose metabolism signaling pathways. Analysis of their expression could help us to understand the possible links between insulin resistance and thyroid nodule.

CONTACTS AND LOCATIONS:
Overall Officials: Fritz-Line FLV VELAYOUDOM, MD, Study Director — CHU de la Guadeloupe
Locations (4):
- France (2):
  - CHU Bordeaux, Bordeaux
  - CHU Limoges, Limoges
- University Hospital Center of Guadeloupe, Pointe-à-Pitre, Guadeloupe
- CHU de la Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anil C, Akkurt A, Ayturk S, Kut A, Gursoy A. Impaired glucose metabolism is a risk factor for increased thyroid volume and nodule prevalence in a mild-to-moderate iodine deficient area. Metabolism. 2013 Jul;62(7):970-5. doi: 10.1016/j.metabol.2013.01.009. Epub 2013 Feb 5. PMID 23395200
- [Background] Ayturk S, Gursoy A, Kut A, Anil C, Nar A, Tutuncu NB. Metabolic syndrome and its components are associated with increased thyroid volume and nodule prevalence in a mild-to-moderate iodine-deficient area. Eur J Endocrinol. 2009 Oct;161(4):599-605. doi: 10.1530/EJE-09-0410. Epub 2009 Jul 24. PMID 19633072
- [Background] Barbesino G. Drugs affecting thyroid function. Thyroid. 2010 Jul;20(7):763-70. doi: 10.1089/thy.2010.1635. PMID 20578900
- [Background] Bonnet F, Scheen A. Understanding and overcoming metformin gastrointestinal intolerance. Diabetes Obes Metab. 2017 Apr;19(4):473-481. doi: 10.1111/dom.12854. Epub 2017 Feb 22. PMID 27987248
- [Background] Chen G, Xu S, Renko K, Derwahl M. Metformin inhibits growth of thyroid carcinoma cells, suppresses self-renewal of derived cancer stem cells, and potentiates the effect of chemotherapeutic agents. J Clin Endocrinol Metab. 2012 Apr;97(4):E510-20. doi: 10.1210/jc.2011-1754. Epub 2012 Jan 25. PMID 22278418
- [Background] Clemmons DR. Structural and functional analysis of insulin-like growth factors. Br Med Bull. 1989 Apr;45(2):465-80. doi: 10.1093/oxfordjournals.bmb.a072335. PMID 2480830
- [Background] American Thyroid Association (ATA) Guidelines Taskforce on Thyroid Nodules and Differentiated Thyroid Cancer; Cooper DS, Doherty GM, Haugen BR, Kloos RT, Lee SL, Mandel SJ, Mazzaferri EL, McIver B, Pacini F, Schlumberger M, Sherman SI, Steward DL, Tuttle RM. Revised American Thyroid Association management guidelines for patients with thyroid nodules and differentiated thyroid cancer. Thyroid. 2009 Nov;19(11):1167-214. doi: 10.1089/thy.2009.0110. PMID 19860577
- [Background] Durante C, Costante G, Lucisano G, Bruno R, Meringolo D, Paciaroni A, Puxeddu E, Torlontano M, Tumino S, Attard M, Lamartina L, Nicolucci A, Filetti S. The natural history of benign thyroid nodules. JAMA. 2015 Mar 3;313(9):926-35. doi: 10.1001/jama.2015.0956. PMID 25734734
- [Background] Hazel-Fernandez L, Xu Y, Moretz C, Meah Y, Baltz J, Lian J, Kimball E, Bouchard J. Historical cohort analysis of treatment patterns for patients with type 2 diabetes initiating metformin monotherapy. Curr Med Res Opin. 2015;31(9):1703-16. doi: 10.1185/03007995.2015.1067194. Epub 2015 Aug 27. PMID 26154837
- [Background] Junik R, Kozinski M, Debska-Kozinska K. Thyroid ultrasound in diabetic patients without overt thyroid disease. Acta Radiol. 2006 Sep;47(7):687-91. doi: 10.1080/02841850600806308. PMID 16950706
- [Background] Levy JC, Matthews DR, Hermans MP. Correct homeostasis model assessment (HOMA) evaluation uses the computer program. Diabetes Care. 1998 Dec;21(12):2191-2. doi: 10.2337/diacare.21.12.2191. No abstract available. PMID 9839117
- [Background] Liu MZ, He HY, Luo JQ, He FZ, Chen ZR, Liu YP, Xiang DX, Zhou HH, Zhang W. Drug-induced hyperglycaemia and diabetes: pharmacogenomics perspectives. Arch Pharm Res. 2018 Jul;41(7):725-736. doi: 10.1007/s12272-018-1039-x. Epub 2018 Jun 1. PMID 29858981
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Menendez C, Baldelli R, Camina JP, Escudero B, Peino R, Dieguez C, Casanueva FF. TSH stimulates leptin secretion by a direct effect on adipocytes. J Endocrinol. 2003 Jan;176(1):7-12. doi: 10.1677/joe.0.1760007. PMID 12525244
- [Background] Meng X, Xu S, Chen G, Derwahl M, Liu C. Metformin and thyroid disease. J Endocrinol. 2017 Apr;233(1):R43-R51. doi: 10.1530/JOE-16-0450. Epub 2017 Feb 14. PMID 28196954
- [Background] Pladevall M, Williams LK, Potts LA, Divine G, Xi H, Lafata JE. Clinical outcomes and adherence to medications measured by claims data in patients with diabetes. Diabetes Care. 2004 Dec;27(12):2800-5. doi: 10.2337/diacare.27.12.2800. PMID 15562188
- [Background] Rezzonico JN, Rezzonico M, Pusiol E, Pitoia F, Niepomniszcze H. Increased prevalence of insulin resistance in patients with differentiated thyroid carcinoma. Metab Syndr Relat Disord. 2009 Aug;7(4):375-80. doi: 10.1089/met.2008.0062. PMID 19320560
- [Background] Rezzonico J, Rezzonico M, Pusiol E, Pitoia F, Niepomniszcze H. Introducing the thyroid gland as another victim of the insulin resistance syndrome. Thyroid. 2008 Apr;18(4):461-4. doi: 10.1089/thy.2007.0223. PMID 18346005
- [Background] Sui M, Yu Y, Zhang H, Di H, Liu C, Fan Y. Efficacy of Metformin for Benign Thyroid Nodules in Subjects With Insulin Resistance: A Systematic Review and Meta-Analysis. Front Endocrinol (Lausanne). 2018 Aug 28;9:494. doi: 10.3389/fendo.2018.00494. eCollection 2018. PMID 30233494
- [Background] Tang Y, Yan T, Wang G, Chen Y, Zhu Y, Jiang Z, Yang M, Li C, Li Z, Yu P, Wang S, Zhu N, Ren Q, Ni C. Correlation between Insulin Resistance and Thyroid Nodule in Type 2 Diabetes Mellitus. Int J Endocrinol. 2017;2017:1617458. doi: 10.1155/2017/1617458. Epub 2017 Oct 12. PMID 29158735
- [Background] Vella V, Sciacca L, Pandini G, Mineo R, Squatrito S, Vigneri R, Belfiore A. The IGF system in thyroid cancer: new concepts. Mol Pathol. 2001 Jun;54(3):121-4. doi: 10.1136/mp.54.3.121. PMID 11376121
- [Background] Wemeau JL, Sadoul JL, d'Herbomez M, Monpeyssen H, Tramalloni J, Leteurtre E, Borson-Chazot F, Caron P, Carnaille B, Leger J, Do Cao C, Klein M, Raingeard I, Desailloud R, Leenhardt L; French Society of Endocrinology. [Recommendations of the French Society of Endocrinology for the management of thyroid nodules]. Presse Med. 2011 Sep;40(9 Pt 1):793-826. No abstract available. French. PMID 22232784
- [Background] Yeo Y, Ma SH, Hwang Y, Horn-Ross PL, Hsing A, Lee KE, Park YJ, Park DJ, Yoo KY, Park SK. Diabetes mellitus and risk of thyroid cancer: a meta-analysis. PLoS One. 2014 Jun 13;9(6):e98135. doi: 10.1371/journal.pone.0098135. eCollection 2014. PMID 24927125
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2008 Jan;31 Suppl 1:S55-60. doi: 10.2337/dc08-S055. No abstract available. PMID 18165338